CLINICAL TRIAL: NCT01658332
Title: Circulating Tumor Cells Identification in Advanced Stage Non-small Cell Lung Cancer
Brief Title: Circulating Tumor Cells in Lung Cancer
Acronym: CIRCUBRONCH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unavailability of the investigator due to an overloaded planning
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-A00135-38
Record Dates: First submitted 2012-06-16; First posted 2012-08-07 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Stage IIIB Non Small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
Keywords: lung cancer; circulating tumor cells; prospective; monocentrique trial
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- specific procedure (Experimental): Circulating tumor cells will be search with the Veridex method at inclusion and after the third chimiotherapy
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — 3 tubes (15 ml)

SUMMARY:
TITLE : Circulating tumor cells identification in advanced stage non-small cell lung cancer (CIRCUBRONCH)

BACKGROUND : Circulating tumor cells identification is a new field of research in oncology, and some studies have been conducted with success on breast and prostate cancer. Nearly 80% of lung cancers are diagnosed in an advanced stage (IIIB, and IV). Circulating tumor cells identification and monitoring these cells after treatment could help the clinicians to detect relapse or be a prognostic factor.

PRIMARY OBJECTIVE : Circulating tumor cells identification, and monitoring in advanced stage lung cancers (IIIB and IV).

SECONDARY OBJECTIVES : Predictive value of the monitoring of circulating tumor cells on the therapeutic response. Prognostic value of identification of circulating tumor cells at the time of diagnosis.

STUDY DESIGN : This study is a prospective, monocentrique trial analyzing the identification of circulating tumor cells in stage IIIB, and IV non-small cell lung cancers.

Duration of the inclusions: 54 months.

Duration of the study: 66 months.

PROCEDURES : Detection of circulating tumor cells with CellSearch system (Veridex), and a cut-off of 5 cells/7,5 ml of blood.

SAMPLE SIZE : 200 patients

STATISTICAL ANALYSIS : Detection of circulating tumor cells is predicted in 20% of stage IIIB, and IV non-small cell lung cancers included in this study. The cut-off is 5 circulating tumor cells per 7,5 ml of blood.

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage NSCLC (stages IIIB, and IV) with measurable or evaluable disease at diagnosis.
* Age ≥ 18 years.
* Measurable or evaluable disease according to RECIST criteria.
* Ability to sign informed consent.

Exclusion Criteria:

* Prior cancers within 5 years, except for non-melanoma skin cancers, and in situ cervical cancers.
* Prior chemotherapy, radiation or surgery for lung cancer.
* Inability to comply with study and/or follow-up procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Identification of circulating tumor cells in locally advanced, and metastatic non-small cell lung cancer. | 18 months
  Circulating tumor cells will be search with the Veridex method, and a value per 7.5 f blood will be recorded.

SECONDARY OUTCOMES:
Identification of a cellular profile according to clinical factors (sex,histology, …). | 18 months
  epidemiological,and clinical characteristics of patients with advanced lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Christelle CLEMENT-DUCHENE, MD, Principal Investigator — CHU NANCY
Locations (1):
- Christelle Clement-Duchene, Nancy, France